CLINICAL TRIAL: NCT02761655
Title: A Study of a Memory Intervention to Improve Medicine Adherence in Patients With Mild Cognitive Impairments and Family Caregiver Medication Administration
Brief Title: A Study of a Memory Intervention to Improve MA in PWMCI & FCG MA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yi-Chien Chiu, PhD, Associate Professor, Chang Gung University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: NMRPD1E0811
Record Dates: First submitted 2016-04-19; First posted 2016-05-04 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Dementia
Keywords: Dementia; Medication Adherence; Perspective Memory
MeSH Terms: conditions — Dementia; Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Patients in both experimental and control groups will receive educations on cognitive impairment, dementia, community resources, and related medication as well as health promotion for PWCIs. The teaching material will be derived from the online resources such as Alzheimer Disease International and Taiwan Alzheimer's Disease Association (TADA) and reviewed by the expert panel as well. Written information will be given to both groups (patients and FCGs), which will be suitable to general public and address issues of cognitive impairment and FCG involvement.
- Intervention Group (Experimental): Patients in both experimental and control groups will receive educations on cognitive impairment, dementia, community resources, and related medication as well as health promotion for PWCIs. The teaching material will be derived from the online resources such as Alzheimer Disease International and Taiwan Alzheimer's Disease Association (TADA) and reviewed by the expert panel as well. Written information will be given to both groups (patients and FCGs), which will be suitable to general public and address issues of cognitive impairment and FCG involvement. The intervention group will further receive memory strategies training on encoding and retention, retrieval, as well as execution and monitoring.
  Interventions: Behavioral: Memory Strategies

INTERVENTIONS:
Behavioral: Memory Strategies — Memory strategies on encoding retention, retrieval, execution and monitoring
  Arms: Intervention Group

SUMMARY:
Background and Purpose: Previous studies indicate that baseline cognitive abilities, especially prospective memory (PM) significantly influence medication adherence. However, there are only three qualified intervention studies on adherences in persons with cognitive impairment (PWCIs). In addition, family caregivers (FCGs) are often asked to assist PWCIs in managing their medication but FCGs' medication administration hassles are not intensively investigated. Therefore, the purpose of this project is to test the effectiveness and efficacy of a theoretical-based multifaceted memory intervention on medication administration and quality of life in PWCIs living at home and medication administration hassle of their FCGs.

Study Design: This is a three-year project (2015, 8, 1-2018, 7, 31). The aims of the first-year study are: 1.to develop a multifaceted memory intervention based on the paradigm of prospective memory (PM); 2. to pilot test the feasibility of the multifaceted memory intervention through a small randomized control trial. The aims of the second- to third year study are: 3. to examine the effectiveness and efficacy of the intervention (a randomized control trial). The intervention group will receive a cognitive impairment education, medication adherence and memory strategies training, while the control group will receive only the cognitive impairment education program. The duration of the intervention is one month. There will be 4 data collections (baseline, post-intervention 2 4, 6 months). Sample size estimation for the pilot study is 5 dyads for each group. Sample size for the randomized clinical trial is 84 dyads (42 dyads per group). After the attrition rate (10%) is counted, in total, there will be 200 cases (100 dyads). Implications of this project: This three-year program can help to identify those who may benefit from memory training and assist those who may be incompetent living in community. Also this program will extend the current knowledge of the role of PM playing in medication adherence behavior and its relationships with self awareness as well as everyday decision making among PWCIs. In addition, health related professionals can improve PWCI's quality of care and reduce FCG hassle by applying a theoretical guided practice for memory training.

DETAILED DESCRIPTION:
These dyad participants are given more information and a follow up phone call to schedule a home visit for initial screening(24<MMSE<27). During the home visit, the participants will be given the consent forms and explanation of this project regarding the purpose, length of data collection and the types of measures of this study. Investigator will use the electronic monitoring system (EMS) developed by Professor Heh's lab, Chung Yuan Christian University in the Phase I to monitor the medication adherence behavior and pilot test its agreement with the pill count and the FCG observation diary. Investigator will apply for the compensations for participants for who finish the initial adherence observation (4 weeks) (baseline data collection). Those who are enrolled for the 6 month intervention phase will receive additional compensation if funded.

The research assistants are those who received training in the previous project (MOST 102-2314-B-182-050-MY2) but investigator will recruit a new part-time research assistant, a nursing master student, to receive a one-month training course, including: the purpose of this study, the procedures for recruitment, test battery interview skills, the test battery scoring system, data collection using the EMS, data download from the EMS, and basic statistical techniques. Then the newly trained part-time assistant will go to the participating sites for observing at least three PWCIs, practicing the interview skills with dyads, and familiarize herself with the outpatient clinical operational system. The on-site participant physicians in the memory disorder clinics will receive a written letter to explain the purpose of this project and the eligible criteria for the dyads. These physicians will help investigators to identify eligible dyads, while trained research assistants will implement the intervention and education program. The part-time student assistant is responsible for data collection.

The advantages of investigators team. The PI and most of the co-PIs come from the same research lab-Healthy Aging Research Center, Cognitive and Behavioral Indices Lab, Chang Gung University. This lab targets on populations such as normal older adults and those with dementia and disability. Investigator have developed own assessment tools and platform used to share the data such as the Prospective and Retrospective Memory Questionnaire (PRMQ). In the future, Investigator may share imaging technology. Therefore, investigators team has the advantages of integration of expertise. Interactions between experts will facilitate the progress of this project. Specifically, Dr. Hsu (a neurologist) will provide the clinical utility that ensures formal diagnosis and assessment for PWCIs. The external consultant (a psychologist), Professor Hua, will assist in administering psychometric tests, interpretation of data, and consultation on the content of intervention. Investigator have international collaboration partners such as Professor Jersey Liang from the University of Michigan, USA for longitudinal and experimental data analyses consultation and Dr. Heather Wilkinson from Edinburgh University, UK to focus on the dementia friendly community issues. Investigator hold monthly research meeting in the lab. Finally, the PI has research collaboration with Professor Heh, Chung Yuan Christian University, on the work of interactive mathematic training APP for MCI patients. Based on this foundation, Investigator will continue to develop the EMS in this project.

Phase 1 (1st year) procedures. After the dyads sign on the consented forms, Investigator spend about 3 hours to collect demographic data, test battery and teach the dyads how to move of patient's medication into the EMS box which contains a sensor to record when the container is opened. Investigator tell the dyads that the box can help patients count their medication pills and it must be used in each medication-taking event. Investigator also teach FCGs how to fill out a medication diary with their observation of patients' medication taking behavior. For those who have their own medication organizers, Investigator ask them to move one of their medications into the system for consistent measure. The baseline observation of medication adherence will last 4 weeks to screen out those who do not have adherence problems which are defined as adherence is less than or equal to 90% of the inter-dose interval over this 4-week medication monitoring period. The rationale for this inclusion criterion is that other studies found that using the EMS introduces some novelty that can initially boost adherence. Since the EMS is new to the participants who may experience this novelty, Investigator will adopt this stringent criterion comparing with the general definition of medication adherence >= 80% the inter-dose interval. At the end of 4 weeks, the trained part-time student assistant will down load the medication adherence data and remove the system from the dyad's house. If the PWCIs have multiple medications, Investigator will select only one (prioritizing order: dementia treatment, antipsychotic medicine, antihypertensive medicine). All the participant dyads will take turns to use the EMS system. During the first 6 months of the first year, Investigator will develop the teaching material and a protocol for phase I pilot study.

The intervention procedures in the pilot study consists of 5 stages: (1) initial home visit for baseline data collection; (2) measurement of baseline adherence over 4 weeks; (3) random assignment for eligible participants who sign on the informed consent forms to either intervention group or the educational comparison group; (4) four weekly in-home nurse visit to deliver the intervention or education control to the dyads; (5) adherence monitoring and outcome measures (over a 6 month period).

When the dyad participants are referred by the physicians, they will go through the five-stage procedures to collect baseline data and 4-week adherence data (week 1 to week 4). Then the dyads will be randomly assigned into one of the two conditions. Different trained research assistants will conduct follow-up four-weekly in-home visits (week 5-8) to deliver the intervention or the educational comparison. During the follow-up (week5-8) home visit, research nurses assigned to the intervention group will review the recommended strategies and tailor these strategies based on individual differences and difficulties in implementing the strategies. Problem-solving will be used to help the dyads. This intervention dose is similar to other studies but we include FCGs to participate in this study and control for PWCIs' awareness levels and their medical decision making capacity.

The fidelity of the intervention will be monitored by a PhD student, using a voice recorder on the intervention nurse' interactions with the dyads. Investigator will track the fidelity whether the intervention protocol is followed. Any difference from the intervention protocol will be examined by reviewing the voice records. Fidelity in the education control group will be monitored by the same procedures as well. To prevent loss of 5-month medication adherence after the end of the 1 month intervention phase, a research assistant will conduct home visits of the dyads every 2 months to download the medication adherence data from the EMS and serve as a memory cue to remind the PWCIs to take their medication. This is a strategy consist with investigator's PM theory as well as Insel et al. and may strengthen the multifaceted memory intervention. However, the research assistant(s) making visits will be careful not to discuss the intervention in both education and intervention conditions.

Blindness. To avoid bias, the PI and the part-time student nurse who collect data as well as the participating physicians can be blind to the condition status of the dyads. Investigator will hire two research assistant(s): one to conduct the memory intervention and the other to conduct the education intervention without inference from each other. These procedures can ensure the double blindness in this project.

Feasibility Indicators for the Phase I-pilot study. The feasibility indicators for the pilot study include the recruitment rate (60%), attrition rates (< 20%), and protocol completion rates (>80%) based on investigator's previous research experiences of recruiting PWCIs into a multiple stimulation intervention through leisure activities.

ELIGIBILITY:
Inclusion Criteria:

* Mandarin Chinese, Taiwanese, and Hakka dialect speakers
* Having a primary FCG who is familiar with patient's conditions and has taken care of the patient or supervised a hired caregiver to take care of the patient in the past three monthshaving a primary FCG who is familiar with patient's conditions and has taken care of the patient or supervised a hired caregiver to take care of the patient in the past three months
* MMSE scores between 27 to 24

Exclusion Criteria:

* Acute illnesses, severe depression (Chinese Geriatric Depression Scale, C-GDS > 10)
* Impaired sensory symptoms (hearing loss and severe visual problems)
* Chronic alcohol abuse or use of drugs

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | Baseline and sixth month after initial visit
  Medical adherence change among patients with cognitive impairment (PWCIs) received intervention in the sixth month after initial visit. The outcome will be measure using Electrical Monitoring System (EMS) and Family Caregivers Observation Diary in adherence rate.
Dementia Quality of Life (DQoL) | Baseline and sixth month after initial visit
  Quality of life change among PWCIs received intervention in the sixth month after initial visit. The outcome will be measured using DQoL questionnaire.

SECONDARY OUTCOMES:
Family Caregivers Medication Administration Hassles (FCG-MAH) | Baseline and sixth month after initial visit
  Change of hassles among family caregivers of in managing medication adherence of PWCIs who received intervention in the sixth month after initial visit. The outcome will be measured using FCG-MAH questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chen Chiu, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan Branch, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided